CLINICAL TRIAL: NCT06514807
Title: A Phase III, Single Arm, Multicentre Study to Evaluate the Efficacy and Safety of Ropeginterferon Alfa-2b in Essential Thrombocythaemia Patients Who Are Intolerant or Refractory to or Not Eligible for Other Cytoreductive Treatments
Brief Title: A Study to Evaluate the Efficacy and Safety of Ropeginterferon Alfa-2b in Essential Thrombocythaemia Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROP-ET
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Essential Thrombocythaemia
Keywords: Ropeginterferon alfa-2b; essential thrombocythaemia; intolerant to cytoreductive treatment; refractory to cytoreductive treatment; not eligible for other cytoreductive treatments; JAK2; CALR; MPL mutation status; BESREMi; Thrombocythaemia
MeSH Terms: conditions — Thrombocythemia, Essential; Thrombocytosis

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, multicentre, descriptive study of ropeginterferon alfa-2b in essential thrombocythaemia patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ropeginterferon alfa-2b (tradename BESREMi®) (Experimental): Ropeginterferon alfa-2b (tradename BESREMi®) 250 micrograms/0.5 mL or 500 micrograms/0.5 ml solution for injection in pre-filled pen.
  Ropeginterferon alfa-2b will be administered subcutaneously every 2 weeks at a dose of 125 µg / 250 µg / 500 µg per injection (depends on the optimal disease response) for up to 36 months of treatment.
  Interventions: Drug: Ropeginterferon alfa-2b (BESREMi®)

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b (BESREMi®) — Ropeginterferon alfa-2b 250 micrograms/0.5 mL or 500 micrograms/0.5 ml solution for injection in pre-filled pen.

SUMMARY:
The primary objective of this study is to assess the efficacy of ropeginterferon alfa-2b in patients with ET who need cytoreductive treatment but are intolerant or refractory to, and/or ineligible for cytoreductive treatments approved and available for the treatment of ET (i.e., HU, ANA, BUS, and PB, when they are available and approved for ET treatment).

Ropeginterferon alfa-2b is currently the only interferon authorised as a cytoreductive treatment of a myeloproliferative neoplasm (MPN), and the long-term treatment data from its comprehensive clinical development program show its efficacy in the induction of haematologic remission, resolution of disease-associated symptoms, disease-modifying effect, as well as its favourable safety profile (Gisslinger et al., 2020; Kiladjian et al. 2022).

Available clinical data and experience show that ropeginterferon alfa-2b normalises various haematological parameters, including platelets. In addition, suppression of the malignant clone causing ET may be achieved, at least after long-term treatment, which is expected to possibly defer the onset of, or avoid long-term sequelae of ET.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient and ability for the patient to comply with the requirements of the study.
2. Male or female patients ≥ 18 years old
3. Patients diagnosed with ET according to the World Health Organization (WHO) 2016 criteria (with a bone marrow biopsy test result not more than 5 years old) who need cytoreductive treatment but are intolerant or refractory to, and/or ineligible for all cytoreductive treatments approved for the treatment of ET (i.e., HU, ANA, BUS, and PB1).

   Patients resistant/intolerant to HU must have documented resistance/intolerance as defined by modified ELN criteria (Barosi, et al. 2007), whereby at least one of the following criteria is met:
   1. Platelet count >600 x 109/L at ≥2 g/day (or ≥2.5 g/day if patient body weight >80 kg) or maximally tolerated dose if <2 g/day or at maximum dose per local practice after at least 3 months of HU
   2. Platelet count >400 x 109/L and WBC count <2.5 x 109/L at any dose and any duration of HU
   3. Platelet count >400 x 109/L and haemoglobin (Hb) <10 g/dL at any dose and any duration of HU
   4. Presence of HU-related toxicities at any dose and any duration of therapy (e.g., leg ulcers, mucocutaneous manifestations, pneumonitis, or HU-related fever)

   Patients resistant/intolerant to ANA, BUS, or PB must meet at least one of the following criteria:
   1. Patient designated as non-responder according to the primary efficacy endpoint of this protocol (modified ELN criteria) after at least 3 months of treatment with the recommended dosing defined in SmPC or local practice
   2. Presence of treatment-related toxicities at any dose and any duration of therapy Patients ineligible for HU: with contraindication as defined by locally available HU SmPC or designated as such by investigator due to benefit-risk concerns (e.g., patients with toxic ranges of myelosuppression, teratogenic/leukaemogenic/carcinogenic concerns, male patients of reproductive, age not willing or unable to use an effective method of contraception). Patients ineligible for ANA: with contraindication as defined by locally available ANA SmPC or designated as such by investigator due to benefit-risk concerns (e.g., cardiovascular risk factors, including heart failure, QT prolongation, the risk for progression to myelofibrosis). Patient ineligible for BUS and PB (in countries where BUS or PB is available and approved for treatment of ET): with contraindication as defined by locally available BUS/PB SmPC or designated as such by investigator due to benefit-risk concerns (e.g., teratogenic/leukaemogenic/carcinogenic concerns, male patients of reproductive age not willing or unable to use an effective method of contraception).
4. If a patient received prior cytoreductive treatment for ET, the washout period between the last dose of treatment and the first dose of the study drug must be at least 14 days, or longer. (If the washout period not completed at time of first patients screening, washout may be done after obtaining ICF during the 28-day screening phase).
5. Interferon treatment-naïve
6. Adequate hepatic function defined as bilirubin ≤1.5 x upper limit normal (ULN), international normalised ratio ≤1.5 x ULN, albumin >3.5 g/dL, alanine aminotransferase ≤2.0 x ULN, aspartate aminotransferase ≤2.0 x ULN at screening.
7. Hospital Anxiety and Depression Scale (HADS) score 0-7 on both subscales.
8. Patient with HADS score of 8-10 inclusive on either, or both, of the subscales may be eligible following psychiatric assessment that excludes clinical significance of the observed symptoms in the context of potential treatment with an interferon alfa.

Exclusion Criteria:

1. Any patient requiring a legally authorised representative
2. Any hypersensitivity to IFN-α or to any of the drug excipients
3. Pre-existing thyroid disease, if not in remission or not controlled with conventional treatment
4. Existence of, or history of severe psychiatric disorders, particularly severe depression, suicidal ideation or suicide attempt
5. Severe cardiovascular disease (i.e., uncontrolled hypertension, congestive heart failure (≥ NYHA class 2), serious cardiac arrhythmia, significant coronary artery stenosis, unstable angina) or recent stroke or myocardial infarction or pulmonary hypertension
6. Patients with diabetes mellitus that cannot be effectively controlled by medicinal products
7. History or presence of autoimmune disease (excluding well-controlled Hashimoto's disease)
8. Immunosuppressed transplant recipients
9. Concomitant treatment with telbivudine
10. Decompensated cirrhosis of the liver (Child-Pugh B or C)
11. End stage renal disease (GFR <15 mL/min)
12. Symptomatic splenomegaly (per the investigator's judgement)
13. Patients with any other significant medical conditions that, in the opinion of the Investigator, would compromise the results of the study or may impair compliance with the requirements of the protocol, including but not limited to:

    1. History of any malignancy within 5 years (except Stage 0 chronic lymphocytic leukaemia, basal cell, squamous cell, and superficial melanoma)
    2. Infections with systemic manifestations (e.g., bacterial, fungal, or human immunodeficiency virus [HIV], except hepatitis B [HBV] and/or hepatitis C [HCV], at screening)
    3. Evidence of severe retinopathy (e.g., cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension)
    4. History of alcohol or drug abuse within the last year
14. Use of any investigational drug <4 weeks prior to the first dose of study drug, or ongoing effects/symptoms due to prior administration of any investigational agent
15. HADS score of 11 or higher on either, or both, of the subscales, and /or development or worsening of the clinically significant depression or suicidal thoughts
16. Pregnant patients or breastfeeding patients or females of childbearing potential not willing to comply with contraceptive requirements as described in Section 16.1.4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Durable (for at least 3 months) peripheral blood count remission | At month 12
  PLTs ≤400 x 109/L AND WBC <10 x 109/L
Absence of haemorrhagic or thrombotic events and absence of disease progression* | At month 12
  *Progression is defined as conversion from asymptomatic to symptomatic splenomegaly or clinically relevant progression of spleen size at the Investigator's discretion, respectively.
Absence or Non-progression* in disease-related signs | At month 12
  *Progression is defined as conversion from asymptomatic to symptomatic splenomegaly or clinically relevant progression of spleen size at the Investigator's discretion, respectively.
Durable (for at least 3 months) large symptoms improvement or maintenance of non-progression based on the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)# | At month 12
  # Large symptoms improvement for ET patients is defined as follows:
  * Baseline TSS ≥20: 10-points reduction in TSS
  * Baseline TSS 15-19, inclusive: 5-points reduction in TSS
  * Baseline TSS 10-14, inclusive: TSS decreases to ≤10
  * Baseline TSS <10: TSS stays <10

SECONDARY OUTCOMES:
Response at month 9, 18, 24, 30 and 36 | Month 9, 18, 24, 30 and 36
Longitudinal changes in the ELN response rates over 12 months | up to 36 months
Time to first response (as defined by ELN criteria) | up to 36 months
Duration of first response (as defined by ELN criteria) | up to 36 months
Duration of first durable response (as defined by ELN criteria) | up to 36 months
Time to first peripheral blood count remission response | up to 36 months
Duration of first durable peripheral blood count remission response | up to 36 months
Occurrence of thromboembolic and bleeding events response | up to 36 months
Occurrence of disease progression response | up to 36 months
Symptomatic improvement assessed by EQ-5D-5L questionnaire response | up to 36 months
Symptomatic improvement assessed by the 10-item MPN-SAF TSS | up to 36 months
Change in inflammation markers over time | up to 36 months
Change in CALR, MPL, or JAK2 allelic burden over time | up to 36 months

OTHER OUTCOMES:
Safety endpoints | up to 36 months
  Adverse events (AEs), according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)

CONTACTS AND LOCATIONS:
Locations (36):
- Austria (4):
  - University Hospital Graz, Department of Internal Medicine, Clinical Department of Hematology, Graz, Styria
  - Medical University Innsbruck, Department of Internal Medicine V (Hematology and Oncology), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen Hospital, Department of Internal Medicine I - Hemato-Oncology, Linz, Upper Austria
  - Medical University Vienna, Department of Internal Medicine I, Clinical Department of Hematology and Hemostaseology, Vienna
- Czechia (2):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Kralovske Vinohrady, Clinic of Internal Hematology, Prague
- France (3):
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, Poitiers
  - Saint-Louis Hospital, Department of Adult Hematology, Paris
  - Bordeaux University Hospital, Haut-Leveque Hospital, Pessac
- Germany (6):
  - University Hospital Aachen, Clinic of Oncology, Hematology and Stem Cell Transplantation (Medical Clinic IV), Aachen
  - University Hospital Halle (Saale), Department of Internal Medicine IV - Hematology and Oncology, Halle
  - Hannover Medical School, Clinic for haematology, haemostaseology, oncology and stem cell transplantation, Hanover
  - University Hospital Mannheim, Medical Clinic III, Hematology and Internistic Oncology, Mannheim
  - Johannes Wesling Hospital Minden, Department of Oncology and Hematology, Minden
  - University Hospital Ulm, Center for Internal Medicine, Clinic of Internal Medicine III, Department of Hematology, Oncology, Rheumatology, Infectious Diseases, Ulm
- Greece (2):
  - General Hospital of Athens Alexandra, Therapeutic Clinic, Department of Therapeutics, Athens
  - University General Hospital "Attikon", Athens
- Hungary (2):
  - Semmelweis University, Department of Internal Medicine and Haematology, Division of Hematology, Budapest
  - University of Debrecen Clinical Center, Clinic of Internal Medicine, Department of Hematology, Debrecen
- Italy (5):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - Careggi University Hospital, Department of Hematology, Florence
  - Umberto I Polyclinic of Rome, Rome
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Service of Hematology, Rome
  - University Hospital City of Health and Science of Turin - Hospital Molinette, Complex Structure of Hematology - U, Turin
- Poland (4):
  - University Teaching Centre, Hematology and Transplantology Clinic, Gdansk
  - Pratia Oncology Katowice, Katowice
  - Independent Public Healthcare Facility University Hospital in Krakow, Teaching Unit of the Hematology Department, Krakow
  - Nicolaus Copernicus Provincial Multispecialty Oncology and Traumatology Center in Lodz, Department of Hematooncology with Subdivision of Daytime Chemotherapy, Lodz
- Romania (4):
  - Onco Card Srl, Brasov
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Hematology Department, Cluj-Napoca
  - Fundeni Clinical Institute, Center for Hematology and Bone Marrow Transplantation, Crişan
  - Iasi Regional Institute of Oncology, Department of Hematology, Iași
- Spain (4):
  - University Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic of Barcelona, Department of Hematology, Barcelona
  - University Hospital Ramon y Cajal, Hematology Service, Madrid
  - Morales Meseguer University General Hospital, Murcia

IPD SHARING:
Plan to Share IPD: No